CLINICAL TRIAL: NCT04402008
Title: A Phase 1/2 Dose Finding Study of Poziotinib in Japanese Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Study of Poziotinib in Japanese Patients With NSCLC
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Business decision, not related to safety.
Sponsor: Spectrum Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPI-POZ-104
Record Dates: First submitted 2020-05-21; First posted 2020-05-26 (Actual); Results first posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-05

CONDITIONS: NSCLC
Keywords: EGFR; HER2; Exon 20 insertion mutation
MeSH Terms: interventions — Clinical Trials, Phase I as Topic

STUDY DESIGN:
Intervention Model Description: Phase 1 will have two randomized, parallel dose groups comparing daily dosing and twice daily dosing at 3 dose levels.
  Phase 2 will be a single dose group evaluating the safety and efficacy of the dose determined in Phase 1 in 2 Cohorts. Cohort 1: EGFR exon 20 insertion mutations and Cohort 2: HER2 exon 20 insertion mutations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase 1: Once Daily Dosing (Experimental): Dose finding at 8 mg, 12 mg, or 16 mg of poziotinib once daily in 28-day treatment cycles.
  Interventions: Drug: Poziotinib Once Daily Dosing
- Phase 1: Twice Daily Dosing (Experimental): Dose finding at 4 mg, 6 mg, or 8 mg of poziotinib twice daily in 28-day treatment cycles.
  Interventions: Drug: Poziotinib Twice Daily Dosing
- Phase 2: Once Daily Dosing or Twice Daily Dosing (Experimental): Once Daily or Twice Daily Dosing as determined in Phase 1 in 28-day treatment cycles.
  Cohort 1: EGFR exon 20 insertion mutations
  Cohort 2: HER2 exon 20 insertion mutations
  Interventions: Drug: Poziotinib Once Daily Dosing or Twice Daily Dosing as determined in Phase 1

INTERVENTIONS:
Drug: Poziotinib Once Daily Dosing — The poziotinib drug substance is a hydrochloride salt of poziotinib and is formulated as a tablet for oral administration.
  Arms: Phase 1: Once Daily Dosing
Drug: Poziotinib Twice Daily Dosing — The poziotinib drug substance is a hydrochloride salt of poziotinib and is formulated as a tablet for oral administration.
  Arms: Phase 1: Twice Daily Dosing
Drug: Poziotinib Once Daily Dosing or Twice Daily Dosing as determined in Phase 1 — The poziotinib drug substance is a hydrochloride salt of poziotinib and is formulated as a tablet for oral administration.
  Arms: Phase 2: Once Daily Dosing or Twice Daily Dosing

SUMMARY:
A Phase 1/2, open-label, multicenter study to determine dose, tolerability, safety and efficacy of poziotinib in Japanese patients non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
This is a Phase 1/2, open-label, multicenter study in Japanese patients with locally advanced or metastatic NSCLC. This study will be conducted in two parts. Phase 1 is designed to observe the maximum tolerated dose (MTD) or maximum administered dose (MAD) of poziotinib when administered once daily or twice daily. Phase 2 will evaluate the safety and efficacy of the dose determined in Phase 1. Study participation includes a 30 day screening period, up to 24 months of treatment, and long-term follow-up for a maximum of 24 months after discontinuation of study treatment.

Phase 1 will enroll up to 36 patients into a dose finding study with two parallel, randomized dose groups. Each group will undergo a dose-finding scheme using a 3+3 design with the assessment of dose-limiting toxicities (DLTs) at up to three dose levels. Patients will be randomized into once daily (QD) or twice daily (BID) dose groups. The DLT assessment will be conducted in the first cycle of treatment and therefore, poziotinib dose modifications are not permitted during this cycle. Patients will be hospitalized for the first 2 weeks.

Phase 2 will enroll 40 additional NSCLC patients with epidermal growth factor receptor (EGFR) (20 patients) or human epidermal growth factor 2 (HER2) (20 patients) exon 20 insertion mutations. Efficacy and safety of the dose and dosing regimen determined in Phase 1 will be evaluated. All patients will be treated in 28-day cycles for up to 24 months.

ELIGIBILITY:
Key Inclusion Criteria:

* Patient must be willing and capable of giving written Informed Consent, adhering to dosing and visit schedules, and meeting all study requirements
* Previously treated patient with histologically or cytologically confirmed (archival tissue accepted) locally advanced or metastatic non-small cell lung cancer (NSCLC) and is not a candidate for definitive therapy

  * Phase 1: No test for mutational status is required
  * Phase 2: Documented EGFR or HER2 exon 20 insertion mutations (including duplication mutations) in NSCLC patients
* Prior treatment status:

  * Phase 1: Patient with refractory NSCLC to available standard therapies
  * Phase 2: Progression after at least one systemic therapy for locally advanced or metastatic disease
* Patient has measurable NSCLC disease, as per the Response Evaluation Criteria in Solid Tumors (RECIST, version 1.1). Metastatic lesions in bone, central nervous system (CNS), or in brain cannot be used for target lesions.
* Patient has recovered from prior systemic therapy for metastatic disease to Grade ≤1 for non-hematologic toxicities (except for Grade ≤2 peripheral neuropathy) and has adequate hematologic, hepatic, and renal function at Baseline

Key Exclusion Criteria:

* Patient is concurrently receiving chemotherapy, biologics, immunotherapy for cancer treatment; systemic anti-cancer treatment or investigational treatment should not be used within 2 weeks prior to Cycle 1, Day 1; local radiation therapy for bone pain may be allowed
* Patient has used strong inhibitors/inducers of CYP3A4 and CYP2D6 within 1 month prior to Cycle 1, Day 1
* Patient has had another primary malignancy within 3 years prior to starting study treatment, except for adequately treated basal or squamous cell carcinoma of the skin or cancer of the cervix in situ
* Patient is pregnant or breastfeeding
* Phase 2 : Patient has had previous treatment with poziotinib. The currently approved tyrosine kinase inhibitors (TKIs) that are not considered to be exon 20 insertion-selective are permissible

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-06-23 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-02-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Japan (3):
  - National Cancer Center East, Kashiwa, Chiba
  - Osaka City General Hospital, Miyakojima-ku, Osaka
  - Shizuoka Cancer Center, Sunto District, Shizuoka

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 42 participants were enrolled at multiple investigative sites in Japan from 23 Jun 2020 to 15 Feb 2023.
Pre-assignment Details: Participants took part in Phase 1 (Dose Escalation) and Phase 2 (Efficacy) of the study. Phase 2 was terminated early.
Groups:
- Phase 1: Poziotinib 8 mg QD: Participants received poziotinib 8 milligrams (mg) orally, once daily (QD) in each 28-day treatment cycle.
- Phase 1: Poziotinib 12 mg QD; Phase 2: Poziotinib 12 mg QD: Participants received poziotinib 12 mg orally, QD in each 28-day treatment cycle.
- Phase 1: Poziotinib 16 mg QD: Participants received poziotinib 16 mg orally, QD in each 28-day treatment cycle.
- Phase 1: Poziotinib 4 mg BID: Participants received poziotinib 4 mg orally, twice daily (BID) in each 28-day treatment cycle.
- Phase 1: Poziotinib 6 mg BID: Participants received poziotinib 6 mg orally, BID in each 28-day treatment cycle.
- Phase 1: Poziotinib 8 mg BID: Participants received poziotinib 8 mg orally, BID in each 28-day treatment cycle.
Period: Overall Study
Arm/Group | Phase 1: Poziotinib 8 mg QD | Phase 1: Poziotinib 12 mg QD | Phase 1: Poziotinib 16 mg QD | Phase 1: Poziotinib 4 mg BID | Phase 1: Poziotinib 6 mg BID | Phase 1: Poziotinib 8 mg BID | Phase 2: Poziotinib 12 mg QD
Started | 3 | 3 | 3 | 4 | 6 | 3 | 20
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 3 | 4 | 6 | 3 | 20
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Disease Progression | 3 | 2 | 3 | 3 | 4 | 3 | 10
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Sponsor Decision | 0 | 0 | 0 | 0 | 0 | 0 | 3
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 0 | 2
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 5

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who signed informed consent, enrolled and received at least 1 dose of poziotinib.
Groups:
- Phase 1: Poziotinib 8 mg QD: Participants received poziotinib 8 mg orally, QD in each 28-day treatment cycle.
- Phase 1:Poziotinib 4 mg BID: Participants received poziotinib 4 mg orally, BID in each 28-day treatment cycle.
- Total: Total of all reporting groups
Arm/Group | Phase 1: Poziotinib 8 mg QD | Phase 1: Poziotinib 12 mg QD | Phase 1: Poziotinib 16 mg QD | Phase 1:Poziotinib 4 mg BID | Phase 1: Poziotinib 6 mg BID | Phase 1: Poziotinib 8 mg BID | Phase 2: Poziotinib 12 mg QD | Total
Number analyzed (Participants) | 3 | 3 | 3 | 4 | 6 | 3 | 20 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (15.01) | 58.7 (12.86) | 65.3 (17.79) | 57.8 (15.26) | 60.3 (15.58) | 52.0 (20.07) | 60.9 (10.36) | 60.1 (12.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1 | 1 | 2 | 3 | 14 | 22
  Male | 3 | 2 | 2 | 3 | 4 | 0 | 6 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 3 | 3 | 4 | 6 | 3 | 20 | 42
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 00 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic/ Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Ethnicity: Not Hispanic/ Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Ethnicity: Japanese | 3 | 3 | 3 | 4 | 6 | 3 | 20 | 42

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: DLT was any of the following treatment-related adverse events occurring during Cycle 1, Non-Hematological Toxicity: Grade 3 or higher toxicity except for alopecia; Grade 3 or higher nausea, vomiting, and diarrhea despite medical intervention. Hematological Toxicity: Grade 4 or higher neutropenia for ≥7 days; Febrile neutropenia with a single temperature of >38.3°C or a sustained temperature of ≥38°C; Neutropenic infection: Grade 3 or higher infection accompanying Grade 4 neutropenia; Grade 4 thrombocytopenia or any grade thrombocytopenia requiring platelet transfusion.
Time Frame: Cycle 1 (Day 1-28)
Population: Safety population included all participants who signed informed consent, enrolled, and received at least 1 dose of poziotinib.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1: Poziotinib 4 mg BID: Participants received poziotinib 4 mg orally, BID in each 28-day treatment cycle.
Arm/Group | Phase 1: Poziotinib 8 mg QD | Phase 1: Poziotinib 12 mg QD | Phase 1: Poziotinib 16 mg QD | Phase 1: Poziotinib 4 mg BID | Phase 1: Poziotinib 6 mg BID | Phase 1: Poziotinib 8 mg BID
Number analyzed (Participants) | 3 | 3 | 3 | 4 | 6 | 3
Participants | 0 | 0 | 3 | 0 | 1 | 2

2. Primary Outcome: Phase 2: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants with best response i.e confirmed complete response (CR) and partial response (PR) as assessed by the investigator using local radiology evaluation according to Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1). CR is defined as the disappearance of all target and non-target lesions. Any pathological lymph nodes must have a reduction in the short axis to <10 millimeters (mm). PR is defined as at least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters, in the absence of CR.
Time Frame: Up to 461 days
Population: Data for this outcome measure was not collected and analyzed as planned as the study was terminated due to the sponsor's business decision.
Arm/Group | Phase 2: Poziotinib 12 mg QD
Number analyzed (Participants) | 0

3. Secondary Outcome: Phase 2: Disease Control Rate (DCR)
Description: The percentage of participants who achieve CR, PR, and stable disease (SD) by the best response from the first dose of poziotinib to the end of the study as assessed by the investigator according to RECIST v1.1. CR is defined as the disappearance of all target and non-target lesions. Any pathological lymph nodes must have reduction in short axis to <10 mm. PR is defined as at least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters, in the absence of CR. SD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum diameters while on study.
Time Frame: Up to 461 days
Population: as for outcome 2
Arm/Group | Phase 2: Poziotinib 12 mg QD
Number analyzed (Participants) | 0

4. Secondary Outcome: Phase 2: Duration of Response (DoR)
Description: Duration of response was defined as the time from the date that measurement criteria are first met for CR or PR until the first subsequent date that progressive disease as assessed by the investigator according to RECIST v1.1 or death is documented. CR is defined as the disappearance of all target and non-target lesions. Any pathological lymph nodes must have a reduction in the short axis to <10 mm. PR is defined as at least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters, in the absence of CR. Disease progression is defined as ≥20% increase in the sum of diameters of target lesions, unequivocal progression in non-target lesions, and/or appearance of new lesions.
Time Frame: Up to 461 days
Population: as for outcome 2
Arm/Group | Phase 2: Poziotinib 12 mg QD
Number analyzed (Participants) | 0

5. Secondary Outcome: Phase 2: Progression Free Survival (PFS)
Description: PFS was the number of days from the treatment start date to the date of first documented disease progression or death from any cause. Per RECIST v1.1 for target lesions, PD was defined as ≥20% increase in sum of diameters (SOD) from previous smallest SOD on study, and an absolute increase of ≥5mm.
Time Frame: Up to 461 days
Population: as for outcome 2
Arm/Group | Phase 2: Poziotinib 12 mg QD
Number analyzed (Participants) | 0

6. Secondary Outcome: Phase 1: Plasma Concentration of Poziotinib and M1, M2 Metabolites
Time Frame: Cycle 1, Day 1 and Day 13
Population: as for outcome 2
Arm/Group | Phase 1: Poziotinib 8 mg QD | Phase 1: Poziotinib 12 mg QD | Phase 1: Poziotinib 16 mg QD | Phase 1: Poziotinib 4 mg BID | Phase 1: Poziotinib 6 mg BID | Phase 1: Poziotinib 8 mg BID
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Phase 1 and 2: Percentage of Participants With Treatment Emergent Adverse Events (TEAE)
Description: TEAEs are AEs that occur from the first dose of study treatment until 40 days after the last dose of study treatment. An AE is defined as any untoward medical occurrence in a patient or clinical investigation patient, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Therefore, an AE can be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product.
Time Frame: Up to 40 days after the last dose of the study drug (Up to 461 days)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1: Poziotinib 8 mg QD | Phase 1: Poziotinib 12 mg QD | Phase 1: Poziotinib 16 mg QD | Phase 1: Poziotinib 4 mg BID | Phase 1: Poziotinib 6 mg BID | Phase 1: Poziotinib 8 mg BID | Phase 2: Poziotinib 12 mg QD
Number analyzed (Participants) | 3 | 3 | 3 | 4 | 6 | 3 | 20
percentage of participants | 100 | 100 | 100 | 100 | 100 | 100 | 100

8. Other Pre Specified Outcome: Phase 2: Exploratory - Overall Survival
Description: The number of days from the treatment start date to the date of death due to any cause.
Time Frame: 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 40 days after the last dose of the study drug (Up to 461 days)
Description: All-cause mortality and AEs: Safety population included all participants who signed informed consent, enrolled, and received at least 1 dose of poziotinib.
Groups:
- Phase 1: Poziotinib 8 mg QD: Participants received poziotinib 8 mg orally, QD, in each 28-day treatment cycle.
- Phase 1: Poziotinib 12 mg QD; Phase 2: Poziotinib 12mg QD: Participants received poziotinib 12 mg orally, QD, in each 28-day treatment cycle.
- Phase 1: Poziotinib 16 mg QD: Participants received poziotinib 16 mg orally, QD, in each 28-day treatment cycle.
- Phase 1: Poziotinib 4 mg BID: Participants received poziotinib 4 mg orally, BID, in each 28-day treatment cycle.
- Phase 1: Poziotinib 6 mg BID: Participants received poziotinib 6 mg orally, BID, in each 28-day treatment cycle.
- Phase 1: Poziotinib 8 mg BID: Participants received poziotinib 8 mg orally, BID, in each 28-day treatment cycle.
Arm/Group | Phase 1: Poziotinib 8 mg QD | Phase 1: Poziotinib 12 mg QD | Phase 1: Poziotinib 16 mg QD | Phase 1: Poziotinib 4 mg BID | Phase 1: Poziotinib 6 mg BID | Phase 1: Poziotinib 8 mg BID | Phase 2: Poziotinib 12mg QD
All-Cause Mortality (participants affected / at risk) | 2/3 | 2/3 | 2/3 | 3/4 | 2/6 | 0/3 | 5/20
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/3 | 0/3 | 1/4 | 1/6 | 0/3 | 4/20
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 4/4 | 6/6 | 3/3 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: Poziotinib 8 mg QD (N=3) | Phase 1: Poziotinib 12 mg QD (N=3) | Phase 1: Poziotinib 16 mg QD (N=3) | Phase 1: Poziotinib 4 mg BID (N=4) | Phase 1: Poziotinib 6 mg BID (N=6) | Phase 1: Poziotinib 8 mg BID (N=3) | Phase 2: Poziotinib 12mg QD (N=20)
Amylase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urethritis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: Poziotinib 8 mg QD (N=3) | Phase 1: Poziotinib 12 mg QD (N=3) | Phase 1: Poziotinib 16 mg QD (N=3) | Phase 1: Poziotinib 4 mg BID (N=4) | Phase 1: Poziotinib 6 mg BID (N=6) | Phase 1: Poziotinib 8 mg BID (N=3) | Phase 2: Poziotinib 12mg QD (N=20)
Diarrhoea (Gastrointestinal disorders) | 1 | 3 | 2 | 2 | 5 | 3 | 17
Stomatitis (Gastrointestinal disorders) | 1 | 3 | 3 | 2 | 4 | 3 | 11
Paronychia (Infections and infestations) | 1 | 2 | 1 | 3 | 3 | 2 | 14
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 | 2 | 3 | 3 | 4 | 0 | 10
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 2 | 1 | 2 | 5
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0 | 0 | 3 | 7
Blepharitis (Eye disorders) | 0 | 1 | 1 | 1 | 1 | 0 | 4
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 3 | 2 | 0 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 4
Angular Cheilitis (Gastrointestinal disorders) | 1 | 1 | 0 | 2 | 1 | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 3
Pyrexia (General disorders) | 1 | 1 | 0 | 1 | 0 | 1 | 3
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 3
Malaise (General disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 3
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 3
Skin atrophy (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 3
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 4
Conjunctivitis (Eye disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Skin infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood corticotrophin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cortisol decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dependent rubor (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eye discharge (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eye inflammation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Glossitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Impetigo (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Peroneal nerve palsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Purpura (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash pustular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tinea pedis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
The study was prematurely terminated for business reasons and not related to safety.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-04): https://cdn.clinicaltrials.gov/large-docs/08/NCT04402008/Prot_SAP_000.pdf